CLINICAL TRIAL: NCT04275440
Title: Effects of Caloric Restriction and Exercise on Body Weight, Cardiometabolic Risk Markers, Immune Function, and Intestinal Flora in College Students: a Randomized Controlled Trial
Brief Title: Effects of Caloric Restriction and Exercise on Body Weight, Immune Function, and Intestinal Flora
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Yanna Zhu, Associate Professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: ZDGW[2019]127
Record Dates: First submitted 2020-02-12; First posted 2020-02-19 (Actual); Last update posted 2021-09-22 (Actual); Status verified 2021-09

CONDITIONS: Cardiometabolic Risk; Weight Loss; Immune System; Intestinal Microbiome
Keywords: Caloric Restriction; Exercise; Young Adult
MeSH Terms: conditions — Weight Loss; Motor Activity | interventions — Exercise; Caloric Restriction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Exercise group (Experimental): Participants would be required to take part in an exercise plan, under the instruction and guidance of professional sports teachers.
  Interventions: Behavioral: Exercise
- Caloric restriction group (Experimental): The caloric restriction plan will be designed based on individual basal metabolic rate.
  Interventions: Behavioral: Caloric restriction
- Combined intervention group (Experimental): Participants will receive both exercise and caloric restriction intervention at the same time.
  Interventions: Behavioral: Exercise; Behavioral: Caloric restriction

INTERVENTIONS:
Behavioral: Exercise — Rope-skipping exercise for three times a week (90 minutes each time, and there is a 10 min break after 20 min Rope skipping). Exercise bracelet and smart bracelet would be used to record the energy consumption throughout the study.
  Arms: Combined intervention group; Exercise group
Behavioral: Caloric restriction — 1. In the first two weeks, participants would reduce their daily energy intake to 100% -110% of his or her basal metabolic energy under instruction, and stick to it till the end of the intervention.
  2. According to the dietary recommendation proposed by Chinese government, participants are required to take in cereals, vegetables, fruits, meat and eggs, while minimize the consumption of sugar-sweeten beverages.
  3. Participants are instructed to arrange their three meals according to the recommended energy distribution (3:4:3).
  Arms: Caloric restriction group; Combined intervention group

SUMMARY:
The purpose of this study is to estimate the effects of caloric restriction and exercise on body weight, cardiovascular metabolic markers, immune function, and intestinal flora among college students, as well as the underlying mechanisms.

DETAILED DESCRIPTION:
In recent decades, carbohydrate-centered food pattern has brought worrying negative effects on human health, including increasing incidence of overweight, obesity, and cardiovascular diseases. Animal experiments based on rhesus monkey showed that caloric restriction could prolong their healthy life years, while reports from population-based studies are quite inconclusive. There are some studies reporting that caloric restriction did reduce the risk of cardiovascular disease in those with obesity, while some other cohort studies found that not eating breakfast might increase the risk of coronary heart disease, diabetes and other related diseases. In addition, a number of studies claimed that continuous caloric restriction is associated with the depletion of peripheral immune cells, immune suppression and reduced bone mineral density. In spite of those inconclusive results, on the whole, fasting and caloric restriction in some way do improve the conditions of metabolism, overweight and obesity. Previous studies mostly focused on middle-aged and elderly people, while recent studies in mice show that energy limitation in elderly people could not stop the aging process genetically or metabolically. Therefore, this study aims to estimate the effects of caloric restriction and exercise on body weight, cardiovascular metabolic markers, immune function, and intestinal flora among college students, as well as the underlying mechanisms. A pilot study containing around 40 participants will be conducted firstly to assess the feasibility of this intervention plan.

ELIGIBILITY:
Inclusion Criteria:

1. First and second year undergraduate students in Sun Yat-sen University.
2. BMI≥22 kg/m2.
3. Having the time and volunteering to receive the interventions.

Exclusion Criteria:

1. Currently engaged in other weight-lossing studies.
2. With secondary obesity induced by medicine or other diseases.
3. With high blood pressure, diabetes or other cadiovascular diseases.
4. Contraindication to exercise.

Ages: 18 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 195 (Actual)
Dates: Start 2019-12-06 (Actual); Primary Completion 2020-04-05 (Actual); Study Completion 2020-04-12 (Actual)

PRIMARY OUTCOMES:
Body weight | Baseline (1-2 days before the intervention), right after intervention (8 weeks), 8 weeks after completion of the intervention
  Body weight change of participants

SECONDARY OUTCOMES:
Body composition | Baseline (1-2 days before the intervention), right after intervention (8 weeks), 8 weeks after completion of the intervention
  Skeletal muscle mass and fat mass were measured by body composition analyzers.
Serum lipid levels | Baseline (1-2 days before the intervention), right after intervention (8 weeks), 8 weeks after completion of the intervention
  Serum lipid levels (total cholesterol, low-density lipoprotein cholesterol, high-density lipoprotein cholesterol, triglycerides) were analyzed by the enzymatic method.
Fasting plasma glucose | Baseline (1-2 days before the intervention), right after intervention (8 weeks), 8 weeks after completion of the intervention
  Fasting plasma glucose were analyzed by the glucose oxidase method.
Systolic and diastolic blood pressure | Baseline (1-2 days before the intervention), right after intervention (8 weeks), 8 weeks after completion of the intervention
  Sitting systolic and diastolic blood pressure were measured with a validated mercury sphygmomanometer (model XJ1ID, China) and TZ-1 stethoscope.
Immune inflammation indicators | Baseline (1-2 days before the intervention), right after intervention (8 weeks), 8 weeks after completion of the intervention
  Immune and inflammatory indicators (ICAM-1, CCL2, VCAM-1, IL-6, IL-8, TNF-alpha, Leptin, Tau, BDNF, VEGF) were analyzed using the Luminex Human Magnetic Assay kit.
Intestinal flora | Baseline (1-2 days before the intervention), right after intervention (8 weeks), 8 weeks after completion of the intervention
  To measure the change of intestinal flora by analyzing feces genome 16S rDNA
Change in scores on Behaviour Rating Inventory of Executive Functioning-Adult Version (BRIEF-A) | Baseline (1-2 days before the intervention), right after intervention (8 weeks), 8 weeks after completion of the intervention
  The executive functions were measured by the Behavior Rating Inventory of Executive Function-Adult Version (BRIEF-A) Self-Report Form. Items are rated 1 (never), 2 (sometimes), and 3 (often). There is no range for a total score. Raw scale scores are used to generate T-scores. A reduction in score indicates less impairment.
Circulating metabolome | Baseline (1-2 days before the intervention), right after intervention (8 weeks), 8 weeks after completion of the intervention
  To measure the change of circulating metabolome by LC-MS/MS method.

CONTACTS AND LOCATIONS:
Overall Officials: Yanna Zhu, M.D, Principal Investigator — Sun Yat-sen University
Locations (1):
- Department of Maternal and Child Health and Sun Yat-sen Global Health Institute, School of Public Health and Institute of State Governance, Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No